CLINICAL TRIAL: NCT03672695
Title: An International Phase Ib Multicentre Study to Characterize the Safety and Tolerability of Intravenously Administered S64315, a Selective Mcl-1 Inhibitor, in Combination With Orally Administered Venetoclax, a Selective Bcl-2 Inhibitor in Patients With Acute Myeloid Leukaemia (AML).
Brief Title: Phase I Dose Escalation Study of Intravenously Administered S64315 in Combination With Orally Administered Venetoclax in Patients With Acute Myeloid Leukaemia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CL1-64315-002; 2018-001809-88 (EudraCT Number)
Record Dates: First submitted 2018-09-04; First posted 2018-09-14 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Initial Schedule - S64315 low dose and venetoclax high dose administered in combination (Experimental)
  Interventions: Combination Product: S 64315 (also referred as MIK665) and venetoclax
- Initial Schedule - S64315 medium dose and venetoclax low dose administered in combination (Experimental)
  Interventions: Combination Product: S 64315 (also referred as MIK665) and venetoclax
- Initial Schedule - S64315 medium dose and venetoclax medium dose administered in combination (Experimental)
  Interventions: Combination Product: S 64315 (also referred as MIK665) and venetoclax
- Initial Schedule - S64315 medium dose and venetoclax high dose administered in combination (Experimental)
  Interventions: Combination Product: S 64315 (also referred as MIK665) and venetoclax
- Initial Schedule - S64315 high dose and venetoclax medium dose administered in combination (Experimental)
  Interventions: Combination Product: S 64315 (also referred as MIK665) and venetoclax
- Alternative Schedule - Venetoclax medium dose administered with no S64315 (Experimental)
  Interventions: Combination Product: S 64315 (also referred as MIK665) and venetoclax
- Alternative Schedule - S64315 medium dose and venetoclax medium dose administered in combination (Experimental)
  Interventions: Combination Product: S 64315 (also referred as MIK665) and venetoclax
- Alternative Schedule - S64315 high dose and venetoclax low dose administered in combination (Experimental)
  Interventions: Combination Product: S 64315 (also referred as MIK665) and venetoclax

INTERVENTIONS:
Combination Product: S 64315 (also referred as MIK665) and venetoclax — The treatment combination period can only begin after the planned dose of venetoclax is reached. Depending on the administration dosing schedule, the combination treatment at the planned doses may be preceded by a 2-week Lead-In Dose period of S64315 (fixed dose) during which the patient continues to receive venetoclax daily. Once the planned dose of both drugs is reached the schedule will be a 21-day cycle with a weekly regimen for S64315 and a daily regimen for venetoclax.
  S64315 should be administered 2 to 4 hours after venetoclax intake, via IV infusion. The dose escalation will start at 50 mg once a week and doses up to 250 mg once a week might be explored.
  Venetoclax will be administered orally once a day. The dose escalation will start at 100 mg daily and doses up to 600 mg daily might be explored. Venetoclax must be taken with a meal (ideally during breakfast) in order to avoid reduced efficacy.

SUMMARY:
The purpose of this study is to determine the safety profile, tolerability and the Recommended Phase 2 Dose of the combination S64315 with venetoclax in patients with Acute Myeloid Leukaemia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years;
2. Patients with cytologically confirmed and documented de novo, secondary or therapy-related AML as defined by World Health Organization (WHO) 2016 classification (Arber, 2016), excluding acute promyelocytic leukaemia (APL, French-American British M3 classification):

   * With relapsed or refractory disease without established alternative therapy or
   * Secondary to MDS treated at least by hypomethylating agent and without established alternative therapy or
   * ≥ 65 years not previously treated for AML and who are not candidates for intensive chemotherapy nor candidates for established alternative therapy
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
4. Able to comply with study procedures
5. Adequate renal function within 7 days before the inclusion of the patient defined as:

   • Serum creatinine ≤ 1.5 x ULN (upper normal limit) or calculated creatinine clearance (determined by MDRD) > 50 mL/min/1.73m2
6. Adequate hepatic function within 7 days before the inclusion of the patient defined as:

   * AST and ALT ≤ 1.5 x ULN
   * Total serum bilirubin level ≤ 1.5 x ULN, except for patients with known Gilbert's syndrome, who are excluded if total bilirubin > 3.0 x ULN or direct bilirubin > 1.5 x ULN

Exclusion Criteria:

1. Participant already enrolled and treated in the study
2. Pregnancy, breastfeeding or possibility of becoming pregnant during the study
3. Participation in another interventional study requiring investigational treatment intake at the same time or within 2 weeks or at least 5 halflives (whichever is longer) prior to first dose of IMP (participation in non-interventional registries or epidemiological studies is allowed). In case of biologic agents with a long half life such as CART cells, immune checkpoint antibodies, bispecific antibodies a flat wash-out of 28 days will be acceptable
4. Presence of ≥ CTCAE Grade 2 toxicity (except alopecia of any grade) due to prior cancer therapy, according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE, version 4.03).
5. Known carriers of HIV antibodies
6. Known history of significant liver disease
7. Uncontrolled hepatitis B or C infection
8. Known active acute or chronic pancreatitis
9. History of myocardial infarction (MI), unstable angina pectoris, coronary artery bypass graft (CABG) within 6 months prior to starting study treatment
10. Any factors that could increase the risk of QTc prolongation or risk of arrhythmic events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLTs) | At the end of cycle 1 (each cycle is 21 or 28 days).
Incidence and severity of AEs | Through study completion, an average of 6 months.
Incidence and severity of SAEs | Through study completion, an average of 6 months.
Number of participants with dose interruptions "will be measured and reported in the Outcome Measure results data table. | Through study completion, an average of 6 months.
Number of participants with dose reductions "will be measured and reported in the Outcome Measure results data table. | Through study completion, an average of 6 months.
Dose intensity | Through study completion, an average of 6 months.

SECONDARY OUTCOMES:
Anti-leukemic activity | Through study completion, an average of 6 months.
  Using blood, bone marrow aspirate and medullary biopsy if available according to ELN 2017 criteria
Pharmacokinetic profile of S64315 administered in combination with Venetoclax in plasma: Area Under the Curve (AUC) | From Day 1 of cycle 1 to the end of cycle 2 (each cycle is 21 or 28 days).
Pharmacokinetic profile of S64315 administered in combination with Venetoclax in plasma: Concentration at the end of infusion (Cinf) | From Day 1 of cycle 1 to the end of cycle 2 (each cycle is 21 or 28 days).
Pharmacokinetic profile of S64315 administered in combination with Venetoclax in plasma: terminal half-life (t½z) | From Day 1 of cycle 1 to the end of cycle 2 (each cycle is 21 or 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew WEI, Principal Investigator — The Alfred Hospital, Melbourne, Victoria
Locations (7):
- United States (2):
  - Smilow Cancer Hospital at Yale, New Haven, Connecticut
  - The University of Texas MD Anderson Cancer Center, Houston, TX, Houston, Texas
- Australia (2):
  - Peter MacCallum cancer centrer, Melbourne
  - The Alfred Hospital Department of Haematology, Victoria Park
- France (3):
  - Institut Paoli-Calmettes, Marseille
  - Hopital Saint-Antoine, Paris
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- See also: Link to Lay Summary and Results Summary — https://clinicaltrials.servier.com/trial/an-international-phase-ib-multicentre-study-to-characterize-the-safety-and-tolerability-of-intravenously-administered-s64315-a-selective-mcl-1-inhibitor-in-combination-with-orally-administered-veneto/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/